CLINICAL TRIAL: NCT02019459
Title: Very Low Nicotine Cigarettes in Smokers With Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Jennifer Tidey, Principal Investigator, Brown University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 5U54DA031659-03 (NIH)
Record Dates: First submitted 2013-12-18; First posted 2013-12-24 (Estimated); Last update posted 2018-04-09 (Actual); Status verified 2018-04

CONDITIONS: Tobacco Dependence
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 0.8 mg nicotine with 10.5 mg tar (Active Comparator): SPECTRUM Cigarette: 0.8 (±0.15) mg nicotine yield with 9 (±1.5) mg tar (standard nicotine and tar yields of commercially-available cigarettes; control condition)
  Interventions: Other: standard nicotine content cigarettes
- 0.03 mg nicotine with 9 mg tar (Experimental): SPECTRUM Cigarette: 0.03 mg (± 0.02) nicotine yield with 9 mg (± 1.5) tar
  Interventions: Other: Very low nicotine content cigarettes

INTERVENTIONS:
Other: Very low nicotine content cigarettes
  Arms: 0.03 mg nicotine with 9 mg tar
Other: standard nicotine content cigarettes
  Arms: 0.8 mg nicotine with 10.5 mg tar

SUMMARY:
Smokers with serious mental illness including those with schizophrenia and bipolar disorder infrequently attempt and attain sustained smoking abstinence and have a 25-year shorter lifespan due to smoking-related illness. This study will examine whether reducing the nicotine content of cigarettes to non-addicting levels is a viable method of reducing smoking in smokers with serious mental illness. Smokers will be randomized to one of two experimental conditions: 1) very low nicotine content (VLNC) cigarettes or 2) normal nicotine content (NNC) cigarettes. Participants will be assessed for patterns of tobacco use, biomarkers of exposure, subjective responses (e.g., satisfaction, craving, withdrawal symptoms), psychiatric symptoms, cognitive performance, smoking cue reactivity and smoking topography.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70
* Schizophrenia, schizoaffective disorder or bipolar disorder
* Smoke an average of at least 10 cigarettes per day for at least 1 year
* Breath carbon monoxide (CO) levels >8 ppm (if ≤ 8 ppm, then nicotine (NicAlert) Strip > 2)

Exclusion Criteria:

* Pregnant or nursing
* Seeking treatment for smoking
* Medical contraindications

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2014-11-17 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Number of cigarettes smoked per day | End of 6 week intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Tidey, Ph.D., Principal Investigator — Brown University
Locations (1):
- Brown University, Providence, Rhode Island, United States